CLINICAL TRIAL: NCT01565018
Title: Single-site, Open-label, Randomized, Cross-over Study in Healthy Japanese Subjects to Evaluate the Bioequivalence of Single Dose Rotigotine Transdermal Patch (2 mg/24 h) Comparing 2 Different Formulations
Brief Title: Bioequivalence Study of Rotigotine Transdermal Patch With Two Different Formulations in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PD0002; 2011-004851-38 (EudraCT Number)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Volunteers
Keywords: Rotigotine; Neupro®; Transdermal Patch; Bioequivalence
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A - Treatment B (Experimental): Treatment A: Test; drug product PR 2.2.1
  Treatment B: Reference; drug product PR 2.1.4
  Sequence of two single applications of Rotigotine transdermal patches (PR 2.2.1 first) for 24 hours separated by a Washout Period of 5 days.
  Interventions: Drug: Rotigotine PR 2.1.4; Drug: Rotigotine PR 2.2.1
- Treatment B - Treatment A (Experimental): Treatment B: Reference; drug product PR 2.1.4
  Treatment A: Test; drug product PR 2.2.1
  Sequence of two single applications of Rotigotine transdermal patches (PR 2.1.4 first) for 24 hours separated by a Washout Period of 5 days.
  Interventions: Drug: Rotigotine PR 2.1.4; Drug: Rotigotine PR 2.2.1

INTERVENTIONS:
Drug: Rotigotine PR 2.1.4 — Treatment B: Rotigotine transdermal patch (2 mg/24 h [10 cm^2]). Reference; drug product PR 2.1.4. Single application of 1 patch for 24 hours.
  Other Names: Neupro
Drug: Rotigotine PR 2.2.1 — Treatment A: Rotigotine transdermal patch (2 mg/24 h [10 cm^2]). Test; drug product PR 2.2.1. Single application of 1 patch for 24 hours.
  Other Names: Neupro

SUMMARY:
To investigate and compare the drug amount delivered to the body after each single administration of Rotigotine patch with 2 different formulations in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male and female volunteers with the age between 20 and 55 years old

Exclusion Criteria:

* Subject has participated or is participating in any other clinical studies of investigational drug or another Investigational Medical Product (IMP) within the last 3 months
* Subject is not healthy (eg, taking any drug treatments, excessive amount of alcohol, cigarettes, having any medical or emotional/psychological problems, a drug/alcohol abuse, having abnormal safety parameters)
* Subject has a QTcB (QT interval corrected for Heart Rate [HR] using Bazett´s formula) interval of ≥ 430 ms (≥ 450 ms for females) or any other clinically relevant finding in Electrocardiogram (ECG) at the Eligibility Assessment (EA)
* Subject is having clinically relevant allergy or clinically relevant drug hypersensitivity to any components of the Investigational Medical Product (IMP), or/and having an atopic or eczematous Dermatitis, Psoriasis and/or active skin disease
* Subject has a recent history (within 2 years) of chronic alcohol or drug abuse and has a history of significant skin hypersensitivity to transdermal products, and of an atopic or eczematous Dermatitis, Psoriasis, and/or active skin disease and have a history of suicide attempt, Epilepsy and/or seizures
* Subject has made a blood donation or a comparable blood loss within the last 3 months prior to the Eligibility Assessment (EA)
* Subject is pregnant or nursing

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of unconjugated Rotigotine (Cmax) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
  The value of the maximum plasma concentration is directly obtained from the observed plasma concentration versus time curves.
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration of unconjugated Rotigotine (AUC 0-t) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from zero up to infinity (AUC(0-∞)) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
  The area under the curve extrapolated to infinity is calculated as the sum of AUC(0-t) and a residual part extrapolated to infinite time.
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration normalized by apparent dose (mg) (AUC(0-t) norm (apparent dose)) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration normalized by body weight (kg) (AUC(0-t) norm (BW)) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Area under the plasma concentration-time curve from zero up to infinity normalized by apparent dose (mg) (AUC(0-∞) norm (apparent dose)) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Area under the plasma concentration-time curve from zero up to infinity normalized by body weight (kg) (AUC(0-∞) norm (BW)) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Maximum plasma concentration normalized by apparent dose (Cmax,norm (apparent dose)) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Maximum plasma concentration normalized by body weight (Cmax,norm (BW)) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Time to reach a maximum plasma concentration of unconjugated Rotigotine after patch application (tmax) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Mean residence time (MRT) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Rate constant of elimination (λz) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Terminal half-life (t1/2) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Relative bioavailability calculated based on maximum plasma concentration (fCmax) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Relative bioavailability calculated based on the area under the plasma concentration-time curve (fAUC) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration
Apparent total body clearance (CL/f) | Pharmacokinetic (PK) samples will be taken predose, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h and 48 h after Rotigotine administration

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 1, Neuss, Germany